CLINICAL TRIAL: NCT01715129
Title: A Phase III Single Arm Study to Evaluate the Efficacy, Safety and Local Tolerability of a Subcutaneous 3-month Formulation of Triptorelin Pamoate (11.25 mg) in Patients With Locally Advanced or Metastatic Prostate Cancer
Brief Title: Induction and Maintenance of Castration After Subcutaneous Injections of Triptorelin Pamoate in Patients With Prostate Cancer
Acronym: DKP 3M SC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8-55-52014-200; 2012-001279-35 (EudraCT Number)
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Results first posted 2015-10-28 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 11.25mg (Experimental): 11.25mg, SC on Day 1 and Day 92
  Interventions: Drug: Triptorelin Pamoate 11.25mg

INTERVENTIONS:
Drug: Triptorelin Pamoate 11.25mg

SUMMARY:
Assess the efficacy and safety of Triptorelin pamoate 3M formulation (11.25mg) when administered by subcutaneous route.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven locally advanced or metastatic prostate cancer who are suitable for androgen deprivation therapy
* Male aged ≥18 years old
* Screening testosterone level of >125 ng/dL
* Life expectancy of greater than 12 months in the judgement of the Investigator
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Willing to give signed informed consent freely
* Able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Prior hormonal therapy for prostate cancer
* Prior surgery or radiotherapy of prostate cancer with curative intent unless disease is verified by a rising prostate specific antigen (PSA) concentration on follow up (elevated PSA values on last two tests conducted at least a month apart) and the patient is eligible for androgen deprivation therapy
* Presence or history of any other malignancy except for non melanoma skin cancer adequately treated at least 2 years before study entry
* Painful local bone lesions or spinal lesions which may lead to compression
* History of myocardial infarction, percutaneous coronary intervention, acute coronary syndrome, coronary artery bypass graft, Class III/IV congestive heart failure, cerebrovascular accident, transient ischaemic attack, or limb claudication at rest, within six months prior to start of study treatment and ongoing symptomatic dysrhythmias, unstable angina, uncontrolled hypertension, and untreated atrial or uncontrolled ventricular arrhythmias
* Any condition in opinion of the Investigator, including other active or latent infections, medical or psychiatric conditions, or the presence of laboratory abnormalities, which could confound the ability to interpret data from the study, compromises the objective of the study or places the patient at unacceptable risk if he participates in the study
* Abnormal haematological, hepatic or renal functions:

  * Haemoglobin <9 g/dL, absolute neutrophil count ≤1.5 x 10^9/L or platelets ≤100 x 10^9/L
  * Serum creatinine ≥1.5 times the upper limit of normal (ULN)
  * Aspartate aminotransferase or alanine aminotransferase >2.5 times the ULN
* Known hypersensitivity to the study treatment, to any of its excipients
* Known active use of recreational drug or alcohol dependence in the opinion of the Investigator
* Any current use or use within six months prior to start of treatment, of medications which are known to affect the metabolism and/or secretion of androgenic hormones: e.g. ketoconazole, aminoglutethimide, oestrogens, and progesterone
* Use of systemic corticosteroids (inhaled corticosteroids and topical application of corticosteroids are permitted)
* Aged ≥90 years for the main study and ≥80 years for those included in the pharmacokinetic (PK) patient population
* Participation in any other study or receipt of any investigational compound in the 30 days (or five times the elimination half life if this is longer) prior to study entry
* Any skin or other condition that may preclude s.c. injection administration
* Known brain or epidural metastases.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Uro-Oncology, Study Director — Ipsen
Locations (12):
- Bulgaria (4):
  - Pleven
  - Plovdiv
  - Shumen
  - Varna
- Suresnes, France
- Latvia (2):
  - Daugavpils
  - Riga
- Poland (3):
  - Kutno
  - Warsaw
  - Wroclaw
- Romania (2):
  - Bucharest
  - Craiova

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 139 subjects were screened and 13 subjects were screen failures.
Groups:
- Triptorelin Pamoate: Triptorelin Pamoate corresponding to 11.25 mg of triptorelin administered subcutaneously on Day 1 and 92
Period: Overall Study
Arm/Group | Triptorelin Pamoate
Started | 126
Completed | 117
Not Completed | 9
Not completed — Adverse Event, fatal | 1
Not completed — Lack of Efficacy | 3
Not completed — Protocol Violation | 1
Not completed — Consent Withdrawn | 2
Not completed — Lost to Follow-up | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (7.3)
Sex/Gender, Customized [Number; unit: participants]
  Male | 126
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian / White | 120
  Missing | 6
Height [Mean (Standard Deviation); unit: cm] | 172.2 (6.7)
Weight [Mean (Standard Deviation); unit: kg] | 80.6 (12.8)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 27.16 (3.96)
Prostate Specific Antigen (PSA) [Mean (Standard Deviation); unit: ng/mL] | 133.53 (385.60)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Demonstrating Castration at Day 29 and Maintaining Castration at Day 183
Description: Percentage of subjects castrated (i.e. with serum testosterone <50 ng/dL or 1.735 nmol/L, using the LC-MS/MS method and missing data imputed by immunoassay method (at time points when LC-MS/MS data was planned to be available only) and the proportion with castration maintained at Day 183 (after receiving 2 S.C. administrations of triptorelin pamoate, three months apart); they were calculated along with their respective 95% confidence intervals (CI) using exact methods on the ITT population at Day 29 and on the initially castrated (IC) population at Day 183
Time Frame: At Day 29 and 183
Population: N=Number of subjects attending the visit
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 126
Percentage of subjects
  Day 29 (N=126) | 97.6 [93.2 to 99.5]
  Day 183 (N=119) | 96.6 [91.6 to 99.1]

2. Secondary Outcome: Percentage of Subjects Demonstrating Castration Before Administration of the Second Dose
Description: Percentage of subjects demonstrating castration at Day 92 (before administration of the second dose) were also assessed using the LC-MS/MS method and missing data imputed by immunoassay method (at time points when LC-MS/MS data was planned to be available only) and summarised using descriptive statistics on the ITT and IC populations.
Time Frame: At Day 92
Population: Initially Castrated (IC1) population: All treated subjects with testosterone levels <50 ng/dL at Day 29 or at Day 36, assessed with the LC-MS/MS method and missing data imputed by immunoassay method.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 120
Percentage of subjects | 99.2 [95.4 to 100]

3. Secondary Outcome: Probability of Testosterone <50 ng/dL
Description: Probability of testosterone <50 ng/dL from Day 29 to Day 183 was assessed as a secondary endpoint using the time to event from first administration date to first observed (and subsequently confirmed if assessment not performed at end of study or early withdrawal visits) serum testosterone level ≥50 ng/dL or ≥1.735 nmol/L at or after Day 29, assessed using the LC-MS/MS Method and Missing Data imputed by immunoassay method Kaplan-Meier Analysis.
  LC-MS/MS: Liquid Chromatography-Tandem Mass Spectrometry
Time Frame: Day 29 through Day 183
Population: Intention-to-treat (ITT) population: All treated subjects
Measure: Number (95% Confidence Interval); unit: Proportion of subjects
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 126
Proportion of subjects | 0.96 [0.92 to 0.99]

4. Secondary Outcome: Percentage of Subjects Demonstrating Castration With Testosterone Level <50 ng/dL at Day 95
Description: Percentage of subjects demonstrating castration at Day 95 (3-4 days after administration of the second dose to assess the suppression of acute-on-chronic effect following the second administration) were also assessed using the LC-MS/MS method and missing data imputed by immunoassay method (at time points when LC-MS/MS data was planned to be available only) and summarised using descriptive statistics on the ITT and IC populations.
Time Frame: Day 95
Population: IC1 population.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 119
Percentage of subjects | 98.3 [94.1 to 99.8]

5. Secondary Outcome: Time to Achieve Castration (Tcast)
Description: Time to castration (Tcast) from first administration date until first observed serum testosterone level <50 ng/dL or <1.735 nmol/L evaluated using the immunoassay method only (i.e. defined as the number of days between the injection time at Day 1 and castration achievement)
Time Frame: Up to Day 36
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Day
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 126
Day | 22 [22 to 23]

6. Secondary Outcome: Plasma Triptorelin Levels (Cmin)
Description: Minimal triptorelin plasma concentration at the end of each dosage interval just before the next dose injection (Cmin) for Days 92 and 183 were assessed.
Time Frame: At Day 92 and 183
Population: ITT population. No samples were collected from 4 subjects at Day 92 and 9 subjects at Day 183
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 122
ng/mL
  Day 92 | 0.062 (0.031)
  Day 183 (N=117) | 0.049 (0.027)

7. Secondary Outcome: Percentage Change in Prostate Specific Antigen (PSA) Levels From Baseline in All Subjects
Description: Serum PSA level was presented throughout the study using descriptive statistics displaying raw values, change from Baseline and percentage change from Baseline at each visit in all subjects from the ITT population only. Additionally, the PSA level was described in subjects with elevated PSA levels (i.e. >4 ng/mL) at study entry, and the proportion of subjects with normal PSA levels (i.e. [0-4] ng/mL) at Day 183 compared to Baseline was presented.
Time Frame: From Day 1 (Baseline) to Day 183 (End of study)
Population: ITT population at End of Study (Day 183). One subject had no data.
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 116
Percentage Change | -85.503 (42.410)

8. Secondary Outcome: Percentage of Subjects With Normal and Abnormal PSA Levels at Day 183 (End of Study Visit)
Description: 0-4 ng/mL (normal PSA value)
  >4 ng/mL (abnormal PSA levels)
Time Frame: At Day 183
Population: Subjects completed Day 183 visit (End of Study)
Measure: Number; unit: Percentage of subjects
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 117
Percentage of subjects
  End of Study (0-4 ng/mL) | 84.6
  End of Study (>4 ng/mL) | 15.4

9. Secondary Outcome: Clinically Apparent Tumor Progression
Description: Tumour progression was recorded according to the Investigator's clinical judgement, considering the PSA levels and any other indications of disease; the clinical confirmation might be supplemented by radiological or other investigations or scans if required. The lack of clinically apparent tumour progression was assessed at Day 92 (prior to administration of the second dose) and Day 183 (end of study visit).
Time Frame: Day 92 and 183
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 126
participants
  Day 92: Non Progressive Disease | 122
  Day 92: Progressive Disease | 0
  Day 183: Non Progressive Disease | 114
  Day 183: Progressive Disease | 3

10. Secondary Outcome: Percentage of Subjects With Adverse Events
Time Frame: Up to Day 183
Population: All subjects who received at least one dose of study treatment were included in safety population.
Measure: Number; unit: Percentage of subjects
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 126
Percentage of subjects
  Any Adverse Events | 35.7
  Any Serious Adverse Events (SAEs) | 4.8
  Any Treatment Emergent Adverse Events (TEAEs) | 35.7
  TEAEs Leading to Withdrawal | 0.8
  TEAEs Leading to Death | 0.8
  Maximum Grade NCI-CTC of TEAEs: Grade 5 | 0.8
  Maximum Grade NCI-CTC of TEAEs: Grade 4 | 0
  Maximum Grade NCI-CTC of TEAEs: Grade 3 | 4.0
  Maximum Grade NCI-CTC of TEAEs: Grade 2 | 13.5
  Maximum Grade NCI-CTC of TEAEs: Grade 1 | 27.8
  Most serious causality of TEAEs: Related | 21.4
  Most serious causality of TEAEs: Not related | 26.2

11. Secondary Outcome: Time to Cmax (Tmax) of Triptorelin
Time Frame: At 1, 2, 3, 4, 5, 6, 7, 8 and 24 hours after first dose on Day 1
Population: Pharmacokinetic (PK) profile was assessed in a subset of 18 subjects.
Measure: Median (Full Range); unit: Hours
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 18
Hours | 4.5 [1.01 to 24]

12. Secondary Outcome: Peak Plasma Concentration Value (Cmax) of Triptorelin
Time Frame: At 1, 2, 3, 4, 5, 6, 7, 8 and 24 hours after first dose on Day 1
Population: PK profile was assessed in a subset of 18 subjects.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 18
ng/mL | 18.58 (7.35)

13. Secondary Outcome: Area Under the Concentration Versus Time Curve Between 0 and 24 Hours (AUC0-24) of Triptorelin
Time Frame: At 1, 2, 3, 4, 5, 6, 7, 8 and 24 hours after first dose on Day 1
Population: PK profile was assessed in a subset of 18 subjects.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 18
h*ng/mL | 304.6 (103.7)

14. Secondary Outcome: Cmin of Triptorelin in Subset of 18 Subjects
Time Frame: At Day 92 and 183
Population: Day 92: Four subjects (presenting particularly high levels of triptorelin) were excluded from 18-subject subset.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 18
ng/mL
  Day 92 (N=14) | 0.078 (0.038)
  Day 183 (N=18) | 0.062 (0.023)

ADVERSE EVENTS:
Time Frame: Up to Day 183
Groups:
- Triptorelin Pamoate 11.25 mg: Triptorelin Pamoate corresponding to 11.25 mg of triptorelin administered subcutaneously on Day 1 and 92
Arm/Group | Triptorelin Pamoate 11.25 mg
Serious Adverse Events (participants affected / at risk) | 6/126
Other Adverse Events (participants affected / at risk) | 45/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triptorelin Pamoate 11.25 mg (N=126)
Fibula Fracture (Injury, poisoning and procedural complications) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triptorelin Pamoate 11.25 mg (N=126)
Hot Flush (Vascular disorders) | 13 (13)
Hypertension (Vascular disorders) | 6 (8)
Flushing (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Oedema Peripheral (General disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hyperthermia (General disorders) | 1 (1)
Injection Site Haematoma (General disorders) | 1 (1)
Injection Site Pain (General disorders) | 1 (1)
Injection Site Swelling (General disorders) | 1 (1)
Anger (Psychiatric disorders) | 1 (1)
Nervousness (Psychiatric disorders) | 1 (1)
Erectile Dysfunction (Reproductive system and breast disorders) | 3 (3)
Breast Pain (Reproductive system and breast disorders) | 2 (2)
Breast Swelling (Reproductive system and breast disorders) | 1 (1)
Breast Tenderness (Reproductive system and breast disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Fibula Fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1)
Weight Increased (Investigations) | 12 (12)
Weight Decreased (Investigations) | 7 (7)
Blood Pressure Increased (Investigations) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (2)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (12)
Loss Of Consciousness (Nervous system disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)
Night Sweats (Skin and subcutaneous tissue disorders) | 2 (2)
Hypotrichosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1)
Ear Infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Tooth Abscess (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No